CLINICAL TRIAL: NCT06086366
Title: Presynaptic Imaging in Major Depressive Episodes After COVID-19
Acronym: PCOV
Status: Recruiting | Type: Observational
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Jeff Meyer, Scientist and Head, Neurochemical Imaging Program in Mood and Anxiety Disorders, Brain Health Imaging Centre, Campbell Family Mental Health Research Institute, Centre for Addiction and Mental Health
Other Study IDs: REB#201/2022
Record Dates: First submitted 2023-09-05; First posted 2023-10-17 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Long COVID; Major Depressive Disorder; Major Depressive Episode
Keywords: PET; Long COVID; Major Depressive Disorder; Major Depressive Episode; Anhedonia; Dopamine Neuron Loss
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Depressive Disorder, Major; Anhedonia | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-DNP: Participants that have recovered from mild or moderate COVID-19 respiratory symptoms and have a new onset major depressive episode (MDE).
  Interventions: Other: [11C]DTBZ PET scan; Other: [18F]SDM8 PET scan; Other: MRI scan
- Healthy Control: Participants in good physical health, age- and sex-matched to Group 1 and 2 participants.
  Interventions: Other: [11C]DTBZ PET scan; Other: [18F]SDM8 PET scan; Other: MRI scan

INTERVENTIONS:
Other: [11C]DTBZ PET scan — One [11C]DTBZ scan for vesicular monoamine transporter 2 (VMAT2)
Other: [18F]SDM8 PET scan — One [18F]SDM8 scan for synaptic vesicle glycoprotein 2A (SV2A)
Other: MRI scan — One MRI scan

SUMMARY:
The goal of this observational study focuses on understanding and addressing a subset of persistent neuropsychiatric symptoms occurring within 3 months after mild to moderate COVID-19 infection (COVID-DNP). COVID-DNP encompasses major depressive episodes (MDE) with or without additional neuropsychiatric symptoms.

DETAILED DESCRIPTION:
Participants will undergo two positron emission tomography (PET) scans, one [11C]DTBZ scan (for vesicular monoamine transporter 2 (VMAT2) and one [18F]SDM8 scan (for synaptic vesicle glycoprotein 2A (SV2A)), as well as one magnetic resonance imaging (MRI) scan.

The main question[s] it aims to answer are:

1. The investigators will determine if VMAT2 binding potential (VMAT2 BPND) is reduced in ventral striatum and dorsal putamen in COVID-DNP.
2. The investigators will determine if SV2A total distribution volume (SV2A VT) is reduced in ventral striatum and dorsal putamen in COVID-DNP

ELIGIBILITY:
Inclusion Criteria:

* New onset MDE within 3 months after mild or moderate COVID-19, with MDE verified by the research version SCID for DSM 5. See "Positive COVID-19 diagnosis" listed after inclusion/exclusion criteria for a description of how this is determined.
* Age 18 to 75.
* Good general physical health with no active medical conditions based on self-report (except migraine or PASC).

Exclusion Criteria:

* Use of antidepressants in the previous month (6 weeks for fluoxetine).
* Use of stimulant medication affecting dopamine release in the previous month
* Use of antipsychotics in the previous month
* History of neurological disease (except migraine, and PASC) based on self-report
* Use of medications or herbal products or natural health products with central nervous system effects in past 2 weeks based on self-report
* Presence of cigarette smoking in the past two months, based on self-report
* Lifetime diagnosis of severe Substance or Alcohol Use Disorder, or diagnosis of mild to moderate Substance or Alcohol Use Disorder in the past two years, based on self-report and verified by the Research Version of Structured Clinical Interview for Diagnostic and Statistical Manual-5 (SCID-5-RV)
* Use of recreational drugs, including marijuana, in the past two months, based on self-report and verified by the Research Version of Structured Clinical Interview for Diagnostic and Statistical Manual-5 (SCID-5-RV)
* Positive urine drug or cotinine screen at any timepoint during the study
* History of psychotic symptoms secondary to schizophrenia, schizophreniform, bipolar disorder, or brief psychotic disorder prior to COVID-19, based on self-report and verified by the Research Version of Structured Clinical Interview for Diagnostic and Statistical Manual-5 (SCID-5-RV)
* Currently pregnant, based on self-report or positive pregnancy test at any timepoint during the study, in females (in our PET Centre females up to 65 years of age are given a urine pregnancy test prior to every PET scan)
* Breastfeeding (for females)
* Current disorders of coagulation, blood or ongoing use of anticoagulant medication, based on self-report
* Claustrophobia, based on self-report
* Weight over 400lbs and height over 7ft (requirements for fitting in the scanners and hospital gowns)
* Presence of metal implant, object or electrical devices that are contraindicated for MRI, based on self-report
* Severe allergic reaction to alcohol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recovered from mild to moderate COVID-19 respiratory symptoms with subsequent onset of COVID-DNP
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-08-22 (Actual); Primary Completion 2028-09-10 (Estimated); Study Completion 2028-09-10 (Estimated)

PRIMARY OUTCOMES:
Vesicular Monoamine Transporter 2 Binding Potential (VAMT2 BPND) | within 3 to 4 weeks after initiation of screening
  The investigators will determine if VMAT2 BPND is changed in ventral striatum and dorsal putamen in COVID-DNP.
Synaptic Vesicle Glycoprotein 2A Total Distribution Volume (SV2A VT) | within 3 to 4 weeks after initiation of screening
  The investigators will determine if SV2A VT is changed in ventral striatum and dorsal putamen in COVID-DNP

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Meyer, M.D., PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No